CLINICAL TRIAL: NCT00697762
Title: A Double-Blind Study to Evaluate the Effectiveness and Safety of RWJ-333369 as Adjunctive Therapy in Korean and Japanese Patients With Partial Onset Seizures
Brief Title: Effectiveness and Safety Study for RWJ-333369 as Adjunctive Therapy in Korean and Japanese Patients With Partial Onset Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was stopped based on information from the global phase 3 studies.
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014284; 333369-KJ-02
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Seizures
Keywords: Partial onset seizure; Adjunctive therapy
MeSH Terms: conditions — Seizures | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 003 (Placebo Comparator): Placebo tablet twice daily for 12 weeks
  Interventions: Drug: Placebo
- 002 (Experimental): RWJ-333369 200 mg tablet twice daily for 12 weeks
  Interventions: Drug: RWJ-333369
- 001 (Experimental): RWJ-333369 100 mg tablet twice daily for 12 weeks
  Interventions: Drug: RWJ-333369

INTERVENTIONS:
Drug: RWJ-333369 — 200 mg tablet twice daily for 12 weeks
  Arms: 002
Drug: RWJ-333369 — 100 mg tablet twice daily for 12 weeks
  Arms: 001
Drug: Placebo — Placebo tablet twice daily for 12 weeks
  Arms: 003

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of adjunctive RWJ-333369 at a dose of 200 or 400 mg/day in comparison with placebo in Korean and Japanese partial epilepsy patients who have poor seizure control with one or two antiepileptics (AEDs).

DETAILED DESCRIPTION:
Despite the introduction of new antiepileptic drugs into overseas clinical settings after 1990's, there still exist those patients who cannot control seizures, and thus the advent of newer antiepileptic drugs is being desired. This is a multicenter, placebo-controlled, double-blind (neither the study physician nor the patient knows the name of the study assigned medication), randomized (study drug assigned by chance), parallel-group study. It consists of three periods: Pretreatment Phase (screening and baseline periods), Double-Blind Treatment Phase, and Posttreatment Phase (transitional period or dose-tapering/withdrawal period). Patients who complete Double-Blind Treatment Phase will be qualified to participate in the long-term extension study (Study 333369-KJ-03) following the present study. The primary hypothesis is that at 400mg/day of RWJ-333369 is effective in the adjunctive treatment of patients with partial onset epilepsy, as measured by the percent reduction from baseline in monthly seizure frequency of partial onset seizures. Safety is evaluated based on the following variables; Adverse event, Lab test, Electrocardiogram, Vital signs, Pregnancy test, Physician Withdrawal Checklist. Patients will receive the assigned dose (placebo, 200 mg/day, or 400 mg/day) twice daily orally for 12 weeks (85 days)

ELIGIBILITY:
Inclusion Criteria:

* Body weight of 40 kg or more
* Established diagnosis of partial epilepsy for at least 1 year
* Current treatment with at least one and no more than two antiepileptics (AEDs)
* At least 6 episodes of simple partial motor seizures, complex partial seizures, or secondarily generalized seizures for 2 months (56 days) during the baseline period (No seizure free interval for more than 3 weeks)

Exclusion Criteria:

* Diagnosis of status epilepticus or epilepsia partialis continua within 6 months
* Patients with generalized epileptic syndrome
* Current or previous history of non-epileptic seizures, including psychogenic seizures
* Current or previous history of any serious or medically relevant systemic disease, including clinically apparent hepatic disease, renal failure, malignant neoplasm, insulin-requiring diabetes mellitus, or any disorder
* Patients with clinical evidence of significant cardiac disease
* Current or past (within 1 year) major significant psychotic disorder
* Have an ALT (GPT) greater than 1.5 times the upper reference limit or total bilirubin above the upper reference limit at screening laboratory tests

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Percent reduction in partial seizure frequency (including simple partial motor seizures, complex partial seizures, and secondarily generalized seizures) for Double-Blind Treatment Phase from the baseline period | From begining to end of Double-Blind Treatment Phase (for 12 weeks).

SECONDARY OUTCOMES:
50% responder rate: The proportion of patients with a 50% reduction or more in the number of partial seizures for Double-Blind Treatment Phase from Pretreatment Phase (baseline period) | From begining to end of Double-Blind Treatment Phase (for 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.